CLINICAL TRIAL: NCT07075419
Title: A Phase Ib/II Clinical Trial of JDB153 Combined With Penpulimab for the Treatment of Hepatocellular Carcinoma Refractory to Standard Therapy
Brief Title: JDB153 Combined With Penpulimab for Hepatocellular Carcinoma After Standard Treatment Failure
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Dan Cao, Chief physician, West China Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JDB153-IIT-HCC001
Record Dates: First submitted 2025-07-11; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Refractory Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; JDB153; Penpulimab
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — penpulimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JDB153 (Experimental): Phase Ib Safety Run-in: JDB153 Monotherapy. Initially, 3 patients will be enrolled to receive JDB153 monotherapy for safety and tolerability assessment prior to combination therapy
  Interventions: Drug: JDB153
- JDB153 combined with Penpulimab (Experimental): Combination Treatment Phase: JDB153 + Penpulimab. After completing the JDB153 monotherapy safety assessment, patients will receive combination treatment with JDB153 and Penpulimab
  Interventions: Drug: JDB153; Drug: Penpulimab

INTERVENTIONS:
Drug: JDB153 — JDB153 is administered orally at doses of 600 mg twice daily (1200 mg total daily dose) or 500 mg twice daily (1000 mg total daily dose) based on safety and tolerability assessment.
Drug: Penpulimab — Penpulimab is administered by intravenous infusion at a dose of 200 mg once every 3 weeks (Q3W).
  Arms: JDB153 combined with Penpulimab

SUMMARY:
The goal of this clinical trial is to evaluate the safety and efficacy of JDB153 combined with Penpulimab in patients with hepatocellular carcinoma after standard treatment failure.

DETAILED DESCRIPTION:
This study is a single-arm, single-center, exploratory clinical trial aimed at evaluating the safety and efficacy of JDB153 combined with Penpulimab in patients with hepatocellular carcinoma after standard treatment failure.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed, or clinically diagnosed (according to Primary Liver Cancer 2024 guidelines or American Association for the Study of Liver Diseases [AASLD] hepatocellular carcinoma guidelines) locally advanced unresectable or metastatic hepatocellular carcinoma;
2. Age 18-75 years, inclusive; no sex restrictions;
3. Life expectancy ≥12 weeks;
4. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
5. Documented disease progression following prior standard systemic therapy. For patients who experienced disease progression within 6 months during or after adjuvant chemotherapy, the adjuvant chemotherapy will be considered first-line treatment;
6. Presence of at least one measurable target lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Target lesions must have a maximum diameter of ≥1 cm if identified by helical computed tomography (CT) or ≥2 cm if identified by conventional CT or magnetic resonance imaging (MRI). All imaging must have been performed within 28 days prior to enrollment;
7. Adequate bone marrow and organ function, as evidenced by laboratory test results obtained within 1 week prior to enrollment: Hemoglobin ≥90 g/L; Platelet count ≥75 × 10⁹/L; White blood cell count ≥3.0 × 10⁹/L; Absolute neutrophil count ≥1.5 × 10⁹/L; Total bilirubin ≤1.5 × upper limit of normal (ULN); Serum creatinine ≤1.5 × ULN; Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤5 × ULN. Patients must not have received blood transfusions, granulocyte colony-stimulating factor (G-CSF), or other medical supportive treatments within 14 days prior to study drug administration;
8. Child-Pugh score ≤7;
9. Voluntary participation with provision of written informed consent.

Exclusion Criteria:

1. History of other malignant tumors with disease-free survival <5 years (except cured basal cell carcinoma of the skin, cured cervical carcinoma in situ, and gastrointestinal tumors confirmed to be cured by endoscopic mucosal resection);
2. Previous treatment with penpulimab;
3. Presence of immunodeficiency disease or HIV infection;
4. Severe, uncontrolled acute infection (defined as fever >38°C caused by infection); 5. History of active hepatitis B or active hepatitis C, defined as: HBV DNA titer ≥2000 IU/mL (or 1×10⁴ copies/mL) or HCV RNA ≥lower limit of detection; 6. Severe hepatic or renal dysfunction; or recent history of myocardial infarction (within 3 months); 7. Patients with active or previous autoimmune disease that has the potential for recurrence or poses associated risks (e.g., those who have undergone organ transplantation requiring immunosuppressive therapy). However, patients with Type I diabetes mellitus, hypothyroidism requiring only hormone replacement therapy, or skin diseases not necessitating systemic treatment (e.g., vitiligo, psoriasis, or alopecia) are permitted to enroll; 8. History of interstitial lung disease or non-infectious pneumonitis that is symptomatic or has a history of pulmonary disease that may interfere with the detection or management of suspected drug-related pulmonary toxicity; 9. History of active tuberculosis infection within 1 year prior to first administration of study drug. However, for patients with a history of active tuberculosis infection more than 1 year ago, enrollment is considered appropriate if the investigator determines there is currently no evidence of active tuberculosis; 10. History of chronic diarrhea or presence of complete intestinal obstruction; 11. Patients requiring systemic treatment with corticosteroids (>10 mg/day prednisone equivalent) or other immunosuppressive medications within 14 days prior to administration of study drug. Note: Inhaled or topical steroids, or adrenal replacement therapy (≤10 mg/day prednisone equivalent), are permitted in the absence of active autoimmune disease. Short-term (≤7 days) use of corticosteroids for prophylactic treatment (e.g., contrast media allergy) or for treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reactions caused by contact allergens) is permitted; 12. Concurrent other serious medical or surgical conditions affecting organ function that the investigator considers inappropriate for participation in this clinical trial; 13. Participation in other investigational drug clinical trials within 4 weeks; 14. Pregnant or lactating women, or patients with reproductive potential (men or women who have been post-menopausal for less than 1 year) who are unwilling to use adequate contraceptive measures; 15. Patients with a history of allergic or hypersensitivity reactions to any study drug components; 16. Patients deemed inappropriate for participation in this clinical trial by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Related Adverse Events | Approximately 2 years
  Number of participants experiencing treatment-related adverse events, serious adverse events, dose-limiting toxicities, and adverse events leading to treatment discontinuation, graded according to NCI CTCAE v5.0

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Approximately 2 years
  Proportion of participants achieving complete response (CR) or partial response (PR) according to RECIST v1.1 criteria
Disease Control Rate (DCR) | Approximately 2 years
  Proportion of participants achieving complete response (CR), partial response (PR), or stable disease (SD) according to RECIST v1.1 criteria
Duration of Response (DoR) | Approximately 2 years
  Time from first documented objective response (CR or PR) to disease progression or death from any cause, whichever occurs first, according to RECIST v1.1 criteria
Time to Progression (TTP) | Approximately 2 years
  Time from study enrollment to disease progression according to RECIST v1.1 criteria
Progression-Free Survival (PFS) | Approximately 2 years
  Time from study enrollment to disease progression or death from any cause, whichever occurs first, according to RECIST v1.1 criteria
Overall Survival (OS) | Approximately 2 years
  Time from study enrollment to death from any cause

IPD SHARING:
Plan to Share IPD: No